CLINICAL TRIAL: NCT01212224
Title: Retrospective Safety Study in 12 Months Treatment Nocturia With Minirin Melt in Clinical Practice in Czech Republic
Brief Title: A Study of Minirin Melt in Patients With Nocturia
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE992026 CS37
Record Dates: First submitted 2010-09-21; First posted 2010-09-30 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a confirmation of safety profile for Minirin Melt in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* nocturia

Exclusion Criteria:

* habitual or psychogenic polydipsia
* known or suspected cardiac insufficiency and other conditions requiring treatment with diuretics
* moderate and severe renal insufficiency
* know hyponatremia
* syndrome of inappropriate ADH secretion

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2187 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Verify the safety profile | 12 months

SECONDARY OUTCOMES:
Safety aspect of dosage | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (81):
- Czechia (81):
  - Nemocnice Rudolfa a Stefanie, Benešov
  - Private ambulance Benešov, Benešov
  - Private ambulance Beroun, Beroun
  - Private ambulance - Slezská urologie, s.r.o., Bohumín
  - Health centre Brno, Brno
  - Hospital Accident, Brno
  - Hospital Delta - private ambulance, Brno
  - Private ambulance Uro-Clinic, s.r.o., Brno
  - Urocentrum, Brno
  - Private ambulance, Brno - Zábrdovice
  - Soukromá ambulanc Černošice, Černošice
  - Hospital Česká Lípa, Česká Lípa
  - Hospital Děčín, Děčín
  - Domažlická nemocnice a.s., Domažlice
  - Soukromá ambulance Dvůr Králové, Dvůr Králové
  - Private ambulance, Hanušovice
  - Hospital with health centre, Havířov
  - Hospital Havlíčkův Brod, Havlíčkův Brod
  - Gynekologická ambulance Hluk, Hluk
  - Private ambulance Urologie, s.r.o., Horšovský Týn
  - Hospital Hradec Králové, Hradec Králové
  - Městská nemocnice Hustopeče, Hustopeč U Brna
  - Private ambulance, Jablonec nad Nisou
  - Soukromá ambulance Jablonec nad Nisou, Jablonec nad Nisou
  - Private ambulance, Jilemnice
  - Hospital ambulance, Karlovy Vary
  - Oblastní nemocnice Kladno, Kladno
  - Hospital Krnov, Krnov
  - Hospital Kromeriz, Kroměříž
  - Soukromá ambulance Kuřim, Kuřim
  - Private ambulance, Lanškroun
  - Soukromá ambulance Mohelnice, Mohelnice
  - Hospital Náchod, Náchod
  - Private ambulance, Nový Jičín
  - Hospital Olomouc, Olomouc
  - Private ambulance - Mediol, s.r.o., Olomouc
  - City Hospital, Ostrava
  - Private ambulance, Ostrava - Poruba
  - Vítkovická hospital, Ostrava - Vítkovice
  - Hospital Pelhřimov, Pelhřimov
  - Hospital Plzeň, Pilsen
  - Private ambulance Plzeň, Pilsen
  - Hospital Písek, Písek
  - Private ambulance Prachatice, Prachatice
  - Hospital Bulovka, Prague
  - Hospital Želeniční nemocnice, Prague
  - Medicon, Prague
  - Private ambulance - Urosante s.r.o., Prague
  - Private ambulance Praha 4, Prague
  - Private ambulance Praha 5, Prague
  - Private ambulance, Prague
  - Private gyn. ambulance, Prague
  - Privátní ambulance Dr. A. Antončík, Prague
  - Thomayer Hospital, Prague
  - Urocare, Prague
  - Urocentrum Praha 2, Prague
  - Urology clinic Hospital Praha, Prague
  - Všeobecná fakultní nemocnice, Prague
  - Hospital Přerov, Přerov
  - Private ambulance - Preštice, Přeštice
  - Private ambulance, Rakovník
  - Soukromá ambulance Roudnice nad Labem, Roudnice nad Labem
  - Private ambulance, Rožnov pod Radhoštěm
  - Hospital Řičany - private ambulance, Říčany
  - Soukromá ambulance Štenberk, Štenberk
  - Private ambulance, Šumperk
  - Šumperská nemocnice, Šumperk
  - Hospital Tábor, Tábor
  - Hospital ambulance, Teplice
  - Hospital Třebíč, Třebíč
  - Hospital Podlesí,s.r.o., Třinec
  - Panoch Hospital, Turnov
  - Hospital with health centre, Uherské Hradiště
  - Masaryk Hospital, Ústí nad Labem
  - Hospital Ústí nad Orlicí, Ústí nad Orlicí
  - Nemocnice Valašské Meziříčí, Valašské Meziřící
  - Krajská nemocnice T. Bati, Zlín
  - Medel, s.r.o., Zlín
  - Private ambulance Lékařský dům, Zlín
  - Private ambulance, Zlín
  - UROKAN, s.r.o., Znojmo